CLINICAL TRIAL: NCT04908059
Title: Leukemic Phase of ALK+ Anaplastic Lymphoma in Real-life Practice: Experience of a University Clinical Hematology Laboratory
Brief Title: Leukemic Phase of ALCL
Acronym: LEUK-ALCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8115
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Anaplastic Lymphoma
Keywords: Anaplastic lymphoma; Leukemic phase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collecting data about the rare leukemic presentation of anaplastic lymphoma to study the characteristics of patients with leukemic phase of ALCL

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a leukemic phase of anaplastic lymphoma

Exclusion Criteria:

* None

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting a leukemic phase of anaplastic lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-07-13 (Estimated); Study Completion 2021-07-13 (Estimated)

PRIMARY OUTCOMES:
A retrospective study of the diagnostic description of the leukemic phases of anaplastic lymphoma in real life | Files analysed retrospectively from January 01, 2020 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MAUVIEUX, MD, PhD, Study Director — Hematology Laboratory - Strasbourg University Hospitals
Locations (1):
- Hematology Laboratory - Strasbourg University Hospitals, Strasbourg, France